CLINICAL TRIAL: NCT01591291
Title: 1/2 - Pharmacogenetic Treatments for Alcoholism
Brief Title: Pharmacogenetic Treatments for Alcoholism
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Grant was transferred to University of Maryland and results were reported under NCT02354703.
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G15991
Record Dates: First submitted 2012-04-17; First posted 2012-05-03 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Alcoholism
Keywords: alcohol dependence; alcohol addiction
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron (Experimental)
  Interventions: Drug: Ondansetron + Brief Behavioral Enhancement Treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo + Brief Behavioral Enhancement Treatment

INTERVENTIONS:
Drug: Ondansetron + Brief Behavioral Enhancement Treatment — Ondansetron 4ug/kg twice daily
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebo + Brief Behavioral Enhancement Treatment — Placebo twice daily
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Heavy drinking can cause serious health, family, and economic problems. Finding treatments that are effective in decreasing heavy drinking among alcohol-dependent individuals is, therefore, an important scientific and health goal. A novel and important strategy to enhance alcoholism treatment efforts uses a personalized medicine approach to optimize treatment effects by selecting the "right" patient therapeutically and potentially with a minimum of adverse events, for a specific medication.

This study will extend findings from a randomized double-blind clinical trial of ondansetron, in which the medication was found to reduce drinking among individuals with certain genotypes (i.e., forms of DNA, the material that controls the inheritance of characteristics). The proposed study will address a number of limitations in the prior work, including testing the medication in both European-American and African-American samples.

DETAILED DESCRIPTION:
This study is a 24 week clinical trial. During the 24 weeks participants will receive either ondansetron or placebo. Participants will also receive Brief Behavioral Compliance enhancement Treatment (BBCET) as their psychosocial adjuct weekly in weeks 1 to 12, and then every 2 weeks in weeks 12 to 24. We will enroll two separate population groups (i.e., African-Americans and European-Americans), each with 128 treatment-seeking, alcohol-dependent individuals in a 24-week clinical trial. Subjects in each of these two population groups (N=128/group) will be randomized into 4 cells (N=32/cell) in a 2 (TT vs. TG or GG) × 2 (ondansetron 4 μg/kg twice daily vs. placebo) factorial design. Group assignment will be achieved using a block randomization procedure that balances the treatment groups on PHDD, age, and gender.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent
* Between the ages of 18 and 65 years and weighing within 30% of ideal body weight. Also, patients must weigh at least 40 kg and no more than 155 kg.
* Good physical health as determined by a complete physical examination, an electrocardiogram (EKG) within normal limits, and laboratory screening tests within acceptable parameters.
* Current DSM-IV diagnosis of alcohol dependence
* AUDIT score of ≥8
* Currently drinking ≥14 alcohol units/week for women and ≥21 alcohol units/week for men in the last 30 days, and have met this criteria prior to randomization
* Provide evidence of stable residence in the last month prior to enrollment in the study, and have no plans to move in the next 9 months.
* Literate in English and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments
* Expressed a wish to reduce or stop drinking
* Willingness to participate in behavioral treatments for alcoholism

Exclusion Criteria:

* Please contact site for additional information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Percent heavy drinking days | up to 24 weeks
  The timeline follow-back (TLFB) method of measuring alcohol consumption will be used to get the percent heavy drinking days.

SECONDARY OUTCOMES:
Drinks per drinking day | up to 24 weeks
  From the TLFB data, other measures of drinking such as drinking intensity (drinks per drinking day; DDD) will be derived.
Percentage of days abstinent | up to 24 weeks
  From the TLFB data, other measures of drinking such as the percentage of days abstinent (PDA) will be derived.
Percentage of subjects with no heavy drinking days | up to 24 weeks
  The TLFB will also be used for other experimental measures that we have validated in previous studies, such as the percentage of subjects with no heavy drinking.
Measures of quality of life | Various time points in the study (screen, weeks 1, 4, 8, 12, 16, 20, 24)
  Quality of life will be assessed using the Quality of Life Enjoyment and Satisfaction Questionnaire and Short Index of Problems.
Objective measure of treatment measure and adverse event using RNA | We will collect RNA on screen, weeks 4, 8, 12, 16, 20, 24
  We will collect RNA samples and using genome-wide expression studies of total RNA, we will compare 15 of the most responsive and 15 of the most least responsive on percent heavy drinking days and 15 with the most and 15 with the fewest adverse events, we will identify changes that mediate ondansetron's efficacy and adverse event profile, respestively.

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, DSc, MD, PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Center for Addiction Research and Education, Charlottesville, Virginia
  - University of Virginia Center for Addiction Research and Education, Richmond, Virginia